CLINICAL TRIAL: NCT04001881
Title: The Role of Heart Echocardiography in the Prediction of Spinal-induced Hypotension in Elderly Patients With Reduced Left Ventricular Function.
Brief Title: Echocardiography and Spinal Induced Hypotension.
Status: Completed | Type: Observational
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, THEODOSIOS SARANTEAS, Associate Professor, Attikon Hospital
Other Study IDs: 3332017
Record Dates: First submitted 2019-06-26; First posted 2019-06-28 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Spinal Anesthetic Toxicity
Keywords: inferior vena cava; spinal anesthesia; echocardiography
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypotension group: spinal anesthesia in Hypotensive patients with low LV-EF Transthoracic echocardiography of IVC before spinal anaesthesia
  Interventions: Other: Transthoracic echocardiography; Drug: Spinal anesthesia
- Normotension group: spinal anesthesia IN Normotensive patients with low LV-EF Transthoracic echocardiography of IVC before spinal anaesthesia
  Interventions: Other: Transthoracic echocardiography; Drug: Spinal anesthesia

INTERVENTIONS:
Other: Transthoracic echocardiography — A standard TTE protocol is used in all patients and included the following views: subcostal 4-chamber (SUBC), apical 4-chamber (4CH), apical 2-chamber (2CH), apical 3-chamber (3CH), parasternal long (LAX) and short axis (SAX).
  Other Names: TTE
Drug: Spinal anesthesia — Spinal anesthesia is introduced with a single intrathecal injection of 12 to 18 mg (15 mg average dose) plain ropivacaine (0.75% solution) using a 22 or 25-gauge needle (pencil-point) with the patient in the lateral position.
  Other Names: Neuraxial block

SUMMARY:
Modern guidelines have combined both the maximum diameter of IVC at expiration (dIVC max) and the IVCCI to appreciate right atrial pressure (RAP) measurements and consequently to assess intravascular volume status. In fact, IVC diameter <2.1 cm with IVCCI >20% (quite inspiration) suggests normal RAP of 3mmHg (range, 0-5mmHg), whereas IVC diameter >2.1 cm with IVCCI<20% suggests high RAP of 15mmHg (range, 10-20mmHg). In occasions where the IVC diameter and collapse is not fit the above categories, an intermediate value of 8 mmHg (range, 5-10 mmHg) is applied. From a clinical standpoint, it is conceivable that both measurements must be measured in isolation to enable RAP assessment. To circumvent this limitation the two indices have been consolidated to dIVCmax-to-IVCCI ratio. Although this ratio has been shown high accuracy to predict spinal-induced hypotension in elderly patients with preserved ejection fraction (EF) of the left ventricle (LV), its value in patients with cardiac dysfunction and reduced LV-EF has not been investigated.

From the aforementioned, this study sets out to address the role of dIVCmax-to-IVCCI ratio in the prediction as well as in the management of hypotension after spinal anesthesia in elderly orthopaedic patients with reduced LV-EF.

DETAILED DESCRIPTION:
Methods In the present prospective study, consecutive sampling is been used to recruit elderly patients (age>70 years) hospitalized in the Attikon University Hospital of Athens. Patients is included if they sustain orthopaedic operation of the lower limb under spinal anaesthesia. This study was approved for ethics and consent by the Institutional Review Board/Ethics Committee of the authors' institution.

Patients' medical history, physical examination, ECG, and X-ray assessment are standard practice, supplemented by specific exams or tests (e.g. TTE or pro-BNP levels), are performed per the consultant cardiologist's recommendations. All patients included in our study are American Heart Association/American College of Cardiology(AHA/ACC) stage II or III with ejection fraction (EF) of the left ventricle (LV) between 35 and 50%, and their cardiac disease status always in compensated status; also, patients with right ventricle (RV) dysfunction and severe valvular diseases are not included in the study.

A standard intraoperative TTE protocol is used in all patients and included the following views: subcostal 4-chamber (SUBC), apical 4-chamber (4CH), apical 2-chamber (2CH), apical 3-chamber (3CH), parasternal long (LAX) and short axis (SAX).

All data are saved and stored digitally for off-line, postoperative analysis. The EF is determined using the biplane Simpson's method, by performing automated measurements of LV volumes in 2CH and 4CH views (GE, Auto-EF system).

The LV-EF, stroke volume index (SVI), peripheral vascular resistance (PVR), LV filling pressures (E/Em ratio), right ventricle (RV) function (tricuspid annular plane systolic excursion (TAPSE), tricuspid annular systolic velocity (TASV), fractional area change (FAC), the IVCCI and dIVCmax-to-IVCCI ratio were assessed Stroke volume (SV) and subsequent stroke volume index (SVI=SV/m2) of the LV is assessed by using automated measurements of LV volumes, according to the formula: SV= EDV-ESV, where EDV=end-diastolic LV volume and ESV=end-systolic LV volume. From these data, we also derived values for the assessment of cardiac output (CO =SV x HR), subsequent systemic vascular resistance (SVR =MAP x 80/CO), (mean arterial blood pressure=MAP, HR=heart rate).

IVC measurements include its maximum diameter at the end of expiration (dIVCmax), IVCCI during spontaneous, quiet, breathing, [(IVC maximal diameter - IVC minimal diameter)/IVC maximal diameter] and the ratio (R) of dIVCmax-to-IVCCI; the IVC diameters is measured in the long axis of the IVC and just proximal to the entry of the hepatic veins.

Anesthetic protocol and measurements. Spinal anesthesia is introduced with a single intrathecal injection of 12 to 18 mg (average15 mg plain ropivacaine, 0.75% solution) using a 22 or 25-gauge needle (pencil-point) with the patient in the lateral position. Intraoperative ECG, SPO2 and invasive arterial blood pressure (through an indwelling radial artery catheter) monitoring is used. Patients who are experiencing a MAP less than or equal to 65 mmHg, or greater than or equal to 25% reduction of its baseline preoperative value were considered hypotensive (duration of low MAP: 30sec, time-period: from spinal anesthesia induction to the end of surgery). Arterial hypotension related to blood transfusion for any reason is not considered in our statistical analysis.

Data analysis:A pilot study of 18 patients revealed a detected area under the ROC curve (AUC) of 0.89 for dIVCmax-to-IVCCI, and for IVCCI 0.74, with rank correlation between the two assays being 0.88 in positive and 0.62 in negative cases. Based on this result, a sample of 40 patients will be required to achieve a power of 80% in order to detect significant difference (at a level 0.05) between dIVCmax-to-IVCCI ratio and IVCCI (MedCalc Software, Mariakerke, Belgium). Quantitative variables and proportions are compared with the student t-test or Mann-Whitney and chi-square tests, respectively. Normality is tested by using the Kolmogorov- Smirnov test. We will assess the area under the receiver operator characteristic curve (AUC-ROC) to evaluate the diagnostic performance of echocardiographic parameters in identifying patients who experience spinal-induced hypotension. The grey zone estimation between two cut-off points will be used for clinical utility reasons.

ELIGIBILITY:
Inclusion Criteria:

Orthopaedic trauma patients Reduced LV-EF (35% <EF<50%) Elderly patients

Exclusion Criteria:

* Patients with right ventricle (RV) dysfunction/patients with LV-EF<35%/
* Severe pulmonary hypertension
* Tachycardia (heart rate > 100 beats/min), atrial fibrillation.
* Patients with tricuspid and mitral regurgitation more than grade 2 and those with more than moderate valvular stenosis were excluded.
* Left ventricular dysynchrony
* TAPSE index<16 and/orTDI-tricuspid annulus<10 cm/sec and/or Fractional Area Shortening<35.

Spinal block below T-12 level Overt intraoperative haemorhage

Ages: 70 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients is included if they sustain orthopaedic operation of the lower limb under spinal anaesthesia.
  Patients' medical history, physical examination, ECG, and X-ray assessment are standard practice, supplemented by specific exams or tests (e.g. TTE or pro-BNP levels), are performed per the consultant cardiologist's recommendations. All patients included in our study were American Heart Association/American College of Cardiology(AHA/ACC) stage II or III with ejection fraction (EF) of the left ventricle (LV) between 35 and 50%, and their cardiac disease status always in compensated status
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
Predictive value of dIVCmax-to-IVCCI ratio | 18 months
  Preoperative performance of the dIVCmax-to-IVCCI ratio The main outcome will be the preoperative performance of the dIVCmax-to-IVCCI ratio to foresee the incidence of hypotension after spinal anesthesia in patients with low LV-EF

CONTACTS AND LOCATIONS:
Overall Officials: THEODOSIOS SARANTEAS, PROFESSOR, Principal Investigator — MEDICAL SCHOOL OF ATHENS, GREECE, EU
Locations (1):
- Department of anesthesia ,ATTIKON UNIVERSITY HOSPITAL OF ATHENS, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Saranteas T, Spiliotaki H, Koliantzaki I, Koutsomanolis D, Kopanaki E, Papadimos T, Kostopanagiotou G. The Utility of Echocardiography for the Prediction of Spinal-Induced Hypotension in Elderly Patients: Inferior Vena Cava Assessment Is a Key Player. J Cardiothorac Vasc Anesth. 2019 Sep;33(9):2421-2427. doi: 10.1053/j.jvca.2019.02.032. Epub 2019 Feb 22. PMID 30904260